CLINICAL TRIAL: NCT04147416
Title: A Multi-center, Open-label, Randomized, Propofol-controlled Study Evaluating the Efficacy and Safety of Intravenous Administration of HSK3486 Injectable Emulsion for Sedation in Intensive Care (ICU) Patients Undergoing Mechanical Ventilation
Brief Title: A Study Evaluating the Efficacy and Safety of HSK3486 for Sedation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSK3486-205
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Sedation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK3486 (Experimental): HSK3486 for Sedation
  Interventions: Drug: HSK3486 0.1-0.2 /0.3 mg / kg group
- Propofol (Active Comparator): Propofol for Sedation
  Interventions: Drug: Propofol 0.5-1.0/1.5 mg/kg group

INTERVENTIONS:
Drug: HSK3486 0.1-0.2 /0.3 mg / kg group — Administered with HSK3486 at a loading dose of 0.1-0.2 mg/kg via intravenous pump. Then HSK3486 shall be administered immediately at an initial maintenance dose of 0.3 mg/kg/h respectively.
  Arms: HSK3486
Drug: Propofol 0.5-1.0/1.5 mg/kg group — Administered with Propofol at a loading dose of 0.5-1.0mg/kg via intravenous pump. Then Propofol shall be administered immediately at an initial maintenance dose of 1.5 mg/kg/h respectively.
  Arms: Propofol

SUMMARY:
This is a multi-center, open-label, randomized, propofol-controlled phase II clinical trial.A total of ICU patients undergoing mechanical ventilation are intended to be enrolled and randomly assigned to HSK3486 group and propofol group in a 2:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who need tracheal intubation for mechanical ventilation and need 6-24 h of sedation after randomization, as anticipated;
2. The target RASS score is between +1 and -2;
3. 18 ≤ age < 80 years old; with no restriction on gender;
4. 18 kg/m2 ≤ BMI ≤ 30 kg/m2;
5. The patients or their family members well understand the purpose and significance of the trial, voluntarily participate in this clinical trial, and sign the informed consent form.

Exclusion Criteria:

1. Patients known to be allergic to eggs, soy products, opioids and their antidotes, and propofol; patients having contraindications to propofol, opioids and their antidotes;
2. Patients having the following medical history or evidence at screening, which may increase sedation/anesthesia risk:

   1. Cardiovascular system: Class III and IV heart failure by New York Heart Association (NYHA), Adams-Stokes syndrome; acute coronary syndrome (ACS) within 6 months prior to screening; bradycardia requiring medications and/or heart rate ≤ 50 beats/min; serious arrhythmia history such as Degree II-III atrioventricular block (excluding patients with pacemakers); acute and chronic myocarditis; systolic pressure ≤ 90 mmHg even when large dose of vasoactive drug (such as norepinephrine ≥ 0.6 μg/kg/min) is used;
   2. Patients with mental disorders (such as schizophrenia, depression, etc.) and cognitive impairment; past abuse history of psychotropics and anesthetics, and long-term use of psychotropics;
   3. Patients with moderate to severe hepatic and renal dysfunctions (liver function: Child-Pugh Grade B and C, scale in Annex 9; renal function: glomerular filtration rate eGFR ≤ 60 mL/(min•1.73 m2) [eGFR is calculated with the Modification of Diet in Renal Disease (MDRD) formula: eGFR = 186 × serum creatinine (SCr)-1.154 × age-0.203 × 0.742 (female)]; patients under dialysis;
   4. Epileptic seizures, convulsions; craniocerebral injury, intracranial hypertension, cerebral aneurysms; Glasgow Coma Score (GCS) ≤ 12 (scale in Annex 6); SOFA > 9 (scale in Annex 7);
   5. Expected survival ≤ 72 h;
3. Laboratory measures at screening period meet the following criteria:

   1. Neutrophil count ≤ 1.0 × 10^9/L;
   2. Platelet count ≤ 50 × 10^9/L;
   3. Hemoglobin ≤ 70 g/L;
4. Pregnant or lactating females; fertile females or males reluctant to receive contraception through the study; any subject planning for pregnancy within 1 month after the study (including male subject);
5. Participated in other drug clinical trials within 1 month prior to screening; Other reasons rendering a subject unsuitable for participation in this study as per the judgment of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-07-03 (Actual)

PRIMARY OUTCOMES:
Mean time to sedation | at day 1
  Defined as the mean time during which the hourly RASS is in the range of +1- -2 during the study treatment

SECONDARY OUTCOMES:
Study drug use | at day 1
  Including the loading dose, maintenance dose, additional dose of HSK3486 and propofol, average unit weight dose per hour of HSK3486 or propofol, total and hourly average numbers of dose adjustments
Minimum maintenance dose | at day 1
  Defined as the minimum dose to maintain the target sedation level (RASS between +1 and -2) of the subject for ≥ 2 h and ≥ 4 h during the administration period
Unit weight dose of remedial drug | at day 1
  Defined as the average hourly unit weight dose of sedatives other than propofol administered for maintaining a target sedation level (RASS between +1 and -2) during the administration period
Unit weight dose of remifentanil | at day 1
  Defined as the average hourly unit weight dose of remifentanil for analgesia during the administration period
Extubation time | at day 1
  Defined as the time from ICU admission to extubation (applicable for subjects who have been intubated before admitted to ICU) or the time from intubation to extubation (applicable for subjects who are intubated after admitted to ICU); for withdrawals, the time of extubation is calculated according to the time of discontinuation; if the extubation does not occur within 24 h of administration, the time of extubation is recorded as 24 h
Recovery time | at day 1
  Defined as the time to recover from sedation status to awaken status (RASS ≥ 0) after drug discontinuation, accurate to the minute; if RASS is ≥ 0 at discontinuation, the recovery time is recorded as 0

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guanzhou, Guangdong, China

REFERENCES:
- [Derived] Liu Y, Zuo L, Li X, Nie Y, Chen C, Liu N, Chen M, Wu J, Guan X. Early sedation using ciprofol for intensive care unit patients requiring mechanical ventilation: a pooled post-hoc analysis of data from phase 2 and phase 3 trials. Ann Intensive Care. 2024 Oct 26;14(1):164. doi: 10.1186/s13613-024-01390-3. PMID 39455495
- [Derived] Liu Y, Yu X, Zhu D, Zeng J, Lin Q, Zang B, Chen C, Liu N, Liu X, Gao W, Guan X. Safety and efficacy of ciprofol vs. propofol for sedation in intensive care unit patients with mechanical ventilation: a multi-center, open label, randomized, phase 2 trial. Chin Med J (Engl). 2022 May 5;135(9):1043-1051. doi: 10.1097/CM9.0000000000001912. PMID 34924506